CLINICAL TRIAL: NCT03013218
Title: A Phase 1, Dose Escalation Study of Evorpacept (ALX148) in Patients With Advanced Solid Tumors and Lymphoma (ASPEN-01)
Brief Title: A Study of Evorpacept (ALX148) in Patients With Advanced Solid Tumors and Lymphoma (ASPEN-01)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ALX Oncology Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AT148001
Record Dates: First submitted 2016-12-15; First posted 2017-01-06 (Estimated); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Metastatic Cancer; Solid Tumor; Advanced Cancer; NonHodgkin Lymphoma
Keywords: Neoplasms; CD47; SIRPα; ALX148; Evorpacept
MeSH Terms: conditions — Neoplasm Metastasis; Lymphoma, Non-Hodgkin; Neoplasms | interventions — ALX148; pembrolizumab; Trastuzumab; Rituximab; Ramucirumab; Paclitaxel; Fluorouracil; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Evorpacept (ALX148) (Experimental): The Part 1 Dose Escalation: Evorpacept (ALX148) infusions will be administered weekly or every two weeks.
  Interventions: Drug: Evorpacept (ALX148)
- Evorpacept (ALX148) + Pembrolizumab (Experimental): The Part 2 Dose Escalation/Expansion: Evorpacept (ALX148) infusions will be administered weekly or every two weeks in combination with pembrolizumab infusions.
  Interventions: Drug: Evorpacept (ALX148); Drug: Pembrolizumab
- Evorpacept (ALX148) + Trastuzumab (Experimental): The Part 2 Dose Escalation/Expansion: Evorpacept (ALX148) infusions will be administered weekly or every two weeks in combination with trastuzumab infusions.
  Interventions: Drug: Evorpacept (ALX148); Drug: Trastuzumab
- Evorpacept (ALX148) + Rituximab (Experimental): The Part 2 Dose Escalation/Expansion: Evorpacept (ALX148) infusions will be administered weekly or every two weeks in combination with rituximab infusions.
  Interventions: Drug: Evorpacept (ALX148); Drug: Rituximab
- Evorpacept (ALX148) + Pembrolizumab + 5FU + Platinum (Experimental): The Part 2 Dose Escalation: Evorpacept (ALX148) infusions will be administered weekly or every two weeks in combination with pembrolizumab + 5FU + platinum infusions.
  Interventions: Drug: Evorpacept (ALX148); Drug: Pembrolizumab; Drug: 5-FU + Cisplatin
- Evorpacept (ALX148) + Trastuzumab + Ramucirumab + Paclitaxel (Experimental): The Part 2 Dose Escalation: Evorpacept (ALX148) infusions will be administered weekly or every two weeks in combination with trastuzumab + ramucirumab + paclitaxel infusions.
  Interventions: Drug: Evorpacept (ALX148); Drug: Trastuzumab; Drug: Ramucirumab + Paclitaxel

INTERVENTIONS:
Drug: Evorpacept (ALX148) — Evorpacept (ALX148)
Drug: Pembrolizumab — Keytruda
  Arms: Evorpacept (ALX148) + Pembrolizumab; Evorpacept (ALX148) + Pembrolizumab + 5FU + Platinum
Drug: Trastuzumab — Herceptin
  Arms: Evorpacept (ALX148) + Trastuzumab; Evorpacept (ALX148) + Trastuzumab + Ramucirumab + Paclitaxel
Drug: Rituximab — Rituxan
  Arms: Evorpacept (ALX148) + Rituximab
Drug: Ramucirumab + Paclitaxel — Standard of care chemotherapy
  Arms: Evorpacept (ALX148) + Trastuzumab + Ramucirumab + Paclitaxel
Drug: 5-FU + Cisplatin — Standard of care chemotherapy
  Arms: Evorpacept (ALX148) + Pembrolizumab + 5FU + Platinum

SUMMARY:
A phase 1, dose escalation study of evorpacept (ALX148) in patients with advanced solid tumors and lymphoma

DETAILED DESCRIPTION:
This phase 1 clinical study (AT148001) is an open-label, multi-center, multiple-dose, dose-escalation, safety, PK, and PD study of evorpacept (ALX148). The phase 1 protocol will have 2 parts: a single agent dose escalation phase (Part 1) and a combination therapy phase (Part 2). Part 2 will include an initial dose escalation portion followed by a dose expansion portion. Approximately 184 adult patients are expected to be enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological diagnosis of advanced/metastatic solid tumor malignancy; or relapsed or refractory Non-Hodgkin lymphoma for whom no standard therapy is available..
* Adequate Bone Marrow Function.
* Adequate Renal & Liver Function.
* Adequate Performance Status

Exclusion Criteria:

* Patients with known symptomatic CNS metastases or lepotomeningeal disease requiring steroids.
* Previous high-dose chemotherapy requiring allogenic stem cell rescue.
* Prior treatment with a CD47 or signal regulatory protein (SIRP) alpha targeting agent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2017-02-03 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2025-07-08 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicities (Number of participants with a DLT) | Up to 28 days
  Number of participants with a DLT

CONTACTS AND LOCATIONS:
Locations (10):
- United States (6):
  - University of Colorado Denver, Denver, Colorado
  - Yale University, New Haven, Connecticut
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - START-Midwest, Grand Rapids, Michigan
  - Seattle Cancer Care Alliance, Seattle, Washington
- South Korea (4):
  - Seoul National University Bundang Hospital, Seongnam
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim TM, Lakhani NJ, Soumerai J, Kamdar M, Gainor JF, Messersmith W, Fanning P, Guan S, Jin F, Forgie A, Wan HI, Pons J, Randolph SS, Kim WS. Evorpacept plus rituximab for the treatment of relapsed or refractory non-Hodgkin lymphoma: results from the phase I ASPEN-01 study. Haematologica. 2025 Sep 1;110(9):2102-2112. doi: 10.3324/haematol.2024.286208. Epub 2025 Apr 10. PMID 40207726
- [Derived] Lakhani NJ, Chow LQM, Gainor JF, LoRusso P, Lee KW, Chung HC, Lee J, Bang YJ, Hodi FS, Kim WS, Santana-Davila R, Fanning P, Squifflet P, Jin F, Kuo TC, Wan HI, Pons J, Randolph SS, Messersmith WA. Evorpacept alone and in combination with pembrolizumab or trastuzumab in patients with advanced solid tumours (ASPEN-01): a first-in-human, open-label, multicentre, phase 1 dose-escalation and dose-expansion study. Lancet Oncol. 2021 Dec;22(12):1740-1751. doi: 10.1016/S1470-2045(21)00584-2. Epub 2021 Nov 15. PMID 34793719